CLINICAL TRIAL: NCT02441530
Title: Vitamin D in the Treatment of Primary Dysmenorrhoea: A Prospective Randomised Controlled Trial
Brief Title: Effectiveness of Vitamin D in Primary Dysmenorrhoea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Seda Ates (Unknown); Osman Sevket (Unknown); Mucize Ozdemir (Unknown); Gulsah Ilhan (Unknown); Yildirim, Zeynep Baysal, M.D. (Individual)
Responsible Party: Principal Investigator, Aysegül Özel, Medical Doctor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BezmialemVU
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Primary Dysmenorrhoea
Keywords: vitamin D
MeSH Terms: interventions — Vitamin D; Vitamin E; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- vitamin D (Experimental): 667 unit of vitamin D once a day ,two days before the expected date of menstruation and continued through the first three days of bleeding.
  Interventions: Dietary Supplement: Vitamin D
- vitamin E (Experimental): 200 unit of vitamin E once a day ,two days before the expected date of menstruation and continued through the first three days of bleeding.
  Interventions: Dietary Supplement: Vitamin E
- ibuprofen (Experimental): 400 mg ibuprofen twice a day, two days before the expected date of menstruation and continued through the first three days of bleeding.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Other Names: Devit-3 damla barcod number 8699525590435 ,DEVA Holding AŞ
  Arms: vitamin D
Dietary Supplement: Vitamin E
  Other Names: Evicap d-alfa-Tokoferol, KOÇAK Farma
  Arms: vitamin E
Drug: Ibuprofen
  Other Names: profen Dinçtaş İlaç
  Arms: ibuprofen

SUMMARY:
Vitamin D in the treatment of primary dysmenorrhoea. Design:Randomised controlled trial. Setting:In a university hospital. Population: 142 women aged 16-35 years. Methods: Patients were treated with 667 unit of vitamin D once a day, 200 unit of vitamin E once a day or 400 mg ibuprofen twice a day,2 days before the date of menstruation and continued through the first 3 days, for 2 months. Main outcome measures: Pain score. Results: Mean VAS of vitamin D group was 4,91, was 6,54 in the vitamin E group and was 4,02 in the ibuprofen group Conclusion:Vitamin D and vitamin E are effective in relieving the pain,but the effect of vitamin D are more prominent

DETAILED DESCRIPTION:
An excessive uterine production of prostaglandins is the pathogenic trigger of dysmenorrhoea. Nonsteroidal anti-inflammatory drugs (NSAIDs) are the currently accepted drugs for the management of this disorder. The capacity for synthesizing vitamin D and the presence of vitamin D receptor in human cycling endometrium have also been demonstrated. Because vitamin D reduces the synthesis of prostaglandins, a beneficial effect of vitamin D for the uterus is possible.Vitamin E inhibits the release of arachidonic acid and the conversion of arachidonic acid to prostaglandin via an action on the enzymes phospholipase A2 and cyclooxygenase.

ELIGIBILITY:
Inclusion Criteria:

1. Women had regular menstrual cycles lasted 21 to 35 days, with menstruation lasting 3 to 7 days;
2. Women had to be in good health and taking no medications including calcium, magnesium, vitamin D and oral contraceptives.
3. Women had not a previous history of gynaecological disease, and a normal pelvic examination were eligible.

Exclusion Criteria:

1) Previous and current use of intrauterine contraceptive devices within the 6 months to enrollment was not permitted

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
pain score ,make a mark on a 10-cm visual analog scale (VAS) | 2 months